CLINICAL TRIAL: NCT03470519
Title: Validation of a Newly Developed Food Frequency Questionnaire to Assess Magnesium Intakes
Brief Title: Magnesium Food Frequency Questionnaire
Acronym: MgFFQ
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Deeptha Sukumar, Dr. Deeptha Sukumar, PhD, Drexel University
Other Study IDs: 1501003336R003
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to develop a quick tool to assess magnesium intakes.

DETAILED DESCRIPTION:
The study aims to develop a quick tool to assess magnesium intakes. Participants will be asked to record a complete dietary intake for 14 consecutive days, the magnesium food frequency questionnaire along with a calcium food frequency questionnaire, and a brief participant data form. Data from the 14 day consecutive food diary will be correlated with the food frequency questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 20-75 years of age
* Fluent in spoken and written English

Exclusion Criteria:

* Unable to report continuous food diary for 14 days
* Medical conditions/medications/supplements affecting metabolism and/or magnesium or calcium status

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men and women ages 20-75 years free of chronic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Magnesium Status | 14 days
  Intake (mg/day)

SECONDARY OUTCOMES:
Calcium Status | 14 days
  Intake (mg/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University Nutrition Sciences Research Lab, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared.